CLINICAL TRIAL: NCT02619409
Title: Evaluation of the Duration of Bupivacaine Spinal Block as the Primary Anesthetic for Orthopedic Procedures With and Without Epinephrine Wash
Brief Title: Evaluation of the Duration of Bupivacaine Spinal Block in Orthopedic Procedures With and Without Epinephrine Wash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Eric Bolin, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00039232
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Arthropathy of Hip; Arthropathy of Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Bupivacaine Only (Placebo Comparator): The bupivacaine only group will receive bupivacaine 0.5% 3cc plus sterile saline 0.1cc.
  Interventions: Drug: Bupivacaine Only
- EPI25 group (Active Comparator): The EPI25 group will receive bupivacaine 0.5% 3cc, epinephrine 1:1000 0.025cc, and sterile saline 0.075cc.
  Interventions: Drug: EPI25
- EPI50 group (Active Comparator): The EPI50 group will receive bupivacaine 0.5% 3cc, epinephrine 1:1000 0.05cc, and sterile saline 0.05cc.
  Interventions: Drug: EPI50 group
- EPI75 group (Active Comparator): The EPI75 group will receive bupivacaine 0.5% 3cc, epinephrine 1:1000 0.075 cc, and sterile saline 0.025%.
  Interventions: Drug: EPI75 group
- EPI100 group (Active Comparator): The EPI100 group will receive bupivacaine 0.5% 3cc, and epinephrine 1:1000 0.1cc
  Interventions: Drug: EPI100 group

INTERVENTIONS:
Drug: Bupivacaine Only — The bupivacaine only group will receive bupivacaine 0.5% 3cc plus sterile saline 0.1cc.
  Arms: Bupivacaine Only
Drug: EPI25 — The EPI25 group will receive bupivacaine 0.5% 3cc, epinephrine 1:1000 0.025cc, and sterile saline 0.075cc.
  Arms: EPI25 group
Drug: EPI50 group — The EPI50 group will receive bupivacaine 0.5% 3cc, epinephrine 1:1000 0.05cc, and sterile saline 0.05cc
  Arms: EPI50 group
Drug: EPI75 group — The EPI75 group will receive bupivacaine 0.5% 3cc, epinephrine 1:1000 0.075cc, and sterile saline 0.025%.
  Arms: EPI75 group
Drug: EPI100 group — The EPI100 group will receive bupivacaine 0.5% 3cc, and epinephrine 1:1000 0.1cc.
  Arms: EPI100 group

SUMMARY:
Bupivacaine spinal is commonly performed as the primary anesthetic for orthopedic procedures. In some cases the duration of the block is inadequate. An epinephrine wash is sometimes performed to prolong the duration of the block. The epinephrine wash may prolong the duration of the block, and if it does, to what extent?

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients scheduled for total hip or knee replacement

Exclusion Criteria:

* Patients taking anticoagulation
* Infection at or near the intended needle insertion site
* Patients with sacral decubitus ulcer at or near the intended needle insertion site aortic stenosis
* Complex spine anatomy
* ASA class greater than III
* Failed SAB as determined by the staff anesthesiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bolin, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Wolla CD, Epperson TI, Woltz EM, Wolf BJ, Bolin ED. Prolongation of spinal duration by escalating doses of intrathecal epinephrine in lower limb arthroplasty. Pain Manag. 2023 Nov;13(11):647-654. doi: 10.2217/pmt-2023-0068. Epub 2023 Nov 15. PMID 37965771

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine Only | EPI25 Group | EPI50 Group | EPI75 Group | EPI100 Group
Started | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Only | EPI25 Group | EPI50 Group | EPI75 Group | EPI100 Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Continuous [Mean (Full Range); unit: years] | 70 [53 to 84] | 63 [50 to 73] | 58 [55 to 77] | 67 [53 to 85] | 59 [28 to 71] | 64 [28 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 2 | 5 | 20
  Male | 1 | 2 | 2 | 4 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 2 | 0 | 7
  White | 3 | 5 | 4 | 4 | 6 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sensory Block
Description: Duration of the sensory block at the T12 dermatome will be assessed in the post operative phase
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bupivacaine Only | EPI25 Group | EPI50 Group | EPI75 Group | EPI100 Group
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 3.41 (1.37) | 2.81 (0.42) | 3.23 (0.72) | 3.12 (0.61) | 3.22 (1.02)

2. Primary Outcome: Duration of Motor Block
Description: (hip felxion) of the non operative leg
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bupivacaine Only | EPI25 Group | EPI50 Group | EPI75 Group | EPI100 Group
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 3.74 (1.13) | 3.36 (0.47) | 3.39 (0.60) | 4.06 (0.98) | 5.20 (1.41)

ADVERSE EVENTS:
Arm/Group | Bupivacaine Only | EPI25 Group | EPI50 Group | EPI75 Group | EPI100 Group
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No